CLINICAL TRIAL: NCT04554238
Title: Effectiveness of Armeo Spring Robotic Therapy in the Function of the Upper Limb of Children With Unilateral Spastic Cerebral Palsy Infiltrated With Botulinum Toxin: Single-blind, Parallel Group Randomized Clinical Trial
Brief Title: Effectiveness of Armeo Spring Robotic Therapy in the Function of the Upper Limb of Children With Unilateral Spastic Cerebral Palsy Infiltrated With Botulinum Toxin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sociedad Pro Ayuda del Niño Lisiado (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SDI2019026
Record Dates: First submitted 2020-08-26; First posted 2020-09-18 (Actual); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Cerebral Palsy; Upper Extremity Paresis
Keywords: Unilateral Cerebral Palsy; Upper extremity function; Armeo spring; Occupational Therapy.
MeSH Terms: conditions — Cerebral Palsy; Paresis | interventions — Occupational Therapy

STUDY DESIGN:
Intervention Model Description: The type of study to be developed corresponds to a parallel group randomized clinical trial (RCT) with a superiority study framework, as it seeks to compare the effectiveness of Armeo spring robotic therapy versus conventional occupational therapy in terms of the functionality of the upper limb of children with hemiparesis infiltrated simultaneously with BTA. The trial phase corresponds to phase III.
Who Masked: Outcomes Assessor
Masking Description: Regarding masking, it is impossible for the treating occupational therapist to be unaware of the treatment to be carried out by the treated patient, just as it is impossible for the patient not to identify the treatment to which they access, therefore, this study is single-blind, considering only who performs the evaluations of the study will not know which group corresponds to the evaluated patient.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Armeo spring group (Experimental): Regarding masking, it is impossible for the treating occupational therapist to be unaware of the treatment to be carried out by the treated patient, just as it is impossible for the patient not to identify the treatment to which they access, therefore, this study is single-blind, considering only who performs the evaluations of the study will not know which group corresponds to the evaluated patient.
  Interventions: Device: Armeo spring
- Occupational Therapy group (Active Comparator): It consists of 5 weeks of intervention, with 3 treatment sessions per week, 40 minutes each time. The patient performs active exercises of the paretic upper limb: bimanual play activities, weight bearing, reaches in various planes of motion that favor shoulder flexion, elbow extension, forearm supination, and dissociated finger movements. In addition to passive mobilizations of the shoulder, elbow and wrist and tactile and proprioceptive sensory stimulation and the use of paretic limbs as support or carrying out prehensions.
  Interventions: Other: Occupational Therapy

INTERVENTIONS:
Device: Armeo spring — Armeo spring is an exoskeleton that allows intensive therapy aimed at upper extremity tasks, which can be regulated according to the anthropometric measurements of the child and the objective of the session. The software contains an extensive library of game-like exercises that are run in a motivating and informative virtual reality training environment, clearly showing the functional task to be performed through immediate feedback in a 3D work space.
  Arms: Armeo spring group
Other: Occupational Therapy — This treatment includes passive stretching exercises, weight bearing, stimulation of protective reactions, muscle strengthening exercises and different types of motivating bimanual games, favoring reaching, grasping, exploration and manipulation.
  Arms: Occupational Therapy group

SUMMARY:
Background: Unilateral spastic cerebral palsy (CP) generates an impact on daily activities, mainly due to the functional limitation of the affected upper limb. The use of technologies such as Armeo spring robotic therapy seeks to improve upper limb mobility through innovative and motivating training that facilitates movement.

Objective: To assess the effectiveness of Armeo spring robotic therapy versus conventional occupational therapy regarding the changes in upper limb functionality of children with unilateral spastic CP infiltrated simultaneously with botulinum toxin A (BTA).

Patients and methods: Randomized clinical trial of parallel groups, in children between 4 and 10 years of age diagnosed with unilateral spastic CP and infiltrates with BTA, who received treatment of conventional occupational therapy (group I) or Armeo spring robotic therapy (group II). The intervention consists of 15 sessions of 40 minutes for 5 weeks, 3 times a week. An initial evaluation is applied with QUEST, ABILHAND-Kids, and MACS, which are re-evaluated at 3 and 6 months.

Hypothesis: Armeo spring robotic therapy will obtain better results than conventional occupational therapy in relation to the functionality of the upper limb at the level of manipulative function, quality of movement of the limb and the performance of daily activities.

Expected results: The results of the QUEST and ABILHAND-Kids dimensions assessed before, after and at follow-up will be the primary outcome. The presence of adverse effects will correspond to secondary outcome.

Benefit and limitations: Direct social contribution for patient's rehabilitation by using technology and a contribution to research to update scientific evidence. Possible limitations could be presence of adverse effects and poor adherence to treatment.

DETAILED DESCRIPTION:
The study will contemplate the description of the clinical characteristics of the patients to intervene (sex, age, locality and Manual Classification of Skills system in children with CP - MACS), and the main results consider the quality upper extremity skills test and the questionnaire of Abilhand-kids. Among the secondary outcomes, the presence of adverse effects and adherence to the intervention will be considered, through the record of attendance at the sessions.In relation to standard operating procedures, no statistical calculation of the sample size will be performed as the entire available population will be covered. All children with spastic unilateral Cerebral Palsy between 4 and 10 years of the year 2018 will be selected at Instituto Teletón in the city of Concepción, Chile. The list of those who have recently been infiltrated with botulinum toxin type A in the upper limb and those who have an indication for admission to treatment will be reviewed. A list will be made with the selected users, assigning the child a number for random selection to a specific study group. The list will be sent to the Subdirección de Investigación - Dirección Médica Nacional of Teletón Chile to maintain the masking.

Participants will be randomly assigned using specialized software to the study group (Armeo) and the control group (conventional therapy) to ensure that each participant has an equal probability of being assigned to either of the two groups. After finishing the Armeo spring group treatment and conventional Occupational Therapy, a post-intervention evaluation will be performed at 3 months and follow-up at 6 months.The data collection will be carried out later, through specific sources: clinical history, interview, evaluation guideline, clinical observation and attendance record. To guarantee the registration procedure, it will be determined that at the end of each evaluation period (initial evaluation, post intervention and follow-up) the evaluator will immediately transfer the information to the database, and it will be verified that it matches the evaluated user through the clinical history number assigned.

The processing and statistical analysis of the data will be coded in an Excel spreadsheet and will be processed using statistical software SPSS v17.0. A normality test will be performed to verify the distribution of the data. According to this result, the corresponding position and dispersion measures will be obtained. To contrast the values of the intragroup variables at the different evaluation times, repeated measures tests will be used and, to evaluate the differences between the study groups, T test or Kruskal Wallis tests will be used, considering a level of significance of 5%. As safety considerations for participants, it is that the treatment will be suspended in the event of the presence of adverse events, for example, skin lesions, pain and fatigue.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Unilateral spastic cerebral palsy
* Botulinum toxin infiltration 3 weeks before start
* Manual Ability Classification scale in level I, II and III

Exclusion Criteria:

* Fixed upper extremity contractures
* Not integrate their affected upper limb into activity.
* Difficult to follow instructions
* Epileptic seizures
* Osteoporosis
* Instability in vital pulmonary or cardiovascular functions

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 23 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline of "Quality of Upper Extremity Skills Test" score at 3 and 6 months post intervention | Before, after the interventions (3 months) and 6 months follow-up
  The Quality Upper Extremity Ability Test (QUEST) assesses the quality of upper extremity function in four domains: dissociated movements, grip, protective extension, and weight-bearing. It was designed to evaluate children with neuromotor dysfunction with spasticity and has been validated in children 18 to 8 years of age.
  The scale presents a specific score for each dimension, which is added, and the final value that is transformed into a final percentage (0-100%). This percentage obtained is the one that is statistically analyzed, understanding that a higher percentage represents a better quality of movement.
  The QUEST allows an evaluation of the quality of the movements of one and two hands in individuals with CP but does not allow an evaluation of the quality of life.

SECONDARY OUTCOMES:
Change from Baseline of "Measure of manual ability for children with upper limb impairments; ABILHAND-kids" score at 3 and 6 months post intervention | Before, after the interventions (3 months) and 6 months follow-up
  The ABILHAND-Kids scale (measure of manual ability for children with upper limb impairments) consists of 21 items, mostly bimanual, rated by the parents. Parents report a better perception of their children's ability than the children themselves.
  On this scale, each task had a numerical assignment according to the difficulty perceived by the father: easy = 1; difficult = 2 and impossible = 3, from which the average was obtained, which was statistically analyzed. It is considered that the decrease in the values corresponds to a perception of a greater number of activities that are easy to carry out by the child.
  ABILHAND-Kids is responsive to detect changes after clinical trials using intensive training in children with unilateral CP. Therefore, this scale is potentially useful for assessing functional status.

OTHER OUTCOMES:
Adherence | Through study completion, an average of 7 months
  A treatment and session calendar will be prepared for each user, which will contain the total number of sessions that the patient must perform. At the end of the study, the percentage of adherence of the patient will be determined, calculating the number of sessions performed divided by the total number of scheduled therapies.
Adverse event | Through study completion, an average of 7 months
  The presence of adverse events in any of the study groups, such as pain, muscle fatigue, shoulder subluxation, among others, will be described.

CONTACTS AND LOCATIONS:
Locations (1):
- Ana Aburto Ojeda, Concepción, Bio Bio, Chile

IPD SHARING:
Plan to Share IPD: No
Not, the information from the database will not be provided, since the tutors signed an authorization to participate and deliver the general results of the research, but authorization is not requested to deliver individual data.

REFERENCES:
- [Background] Rosenbaum P, Paneth N, Leviton A, Goldstein M, Bax M, Damiano D, Dan B, Jacobsson B. A report: the definition and classification of cerebral palsy April 2006. Dev Med Child Neurol Suppl. 2007 Feb;109:8-14. PMID 17370477
- [Background] Klingels K, Demeyere I, Jaspers E, De Cock P, Molenaers G, Boyd R, Feys H. Upper limb impairments and their impact on activity measures in children with unilateral cerebral palsy. Eur J Paediatr Neurol. 2012 Sep;16(5):475-84. doi: 10.1016/j.ejpn.2011.12.008. Epub 2012 Jan 13. PMID 22244966
- [Background] Pierce SR, Daly K, Gallagher KG, Gershkoff AM, Schaumburg SW. Constraint-induced therapy for a child with hemiplegic cerebral palsy: a case report. Arch Phys Med Rehabil. 2002 Oct;83(10):1462-3. doi: 10.1053/apmr.2002.34832. PMID 12370887
- [Background] Brown JK, van Rensburg F, Walsh G, Lakie M, Wright GW. A neurological study of hand function of hemiplegic children. Dev Med Child Neurol. 1987 Jun;29(3):287-304. doi: 10.1111/j.1469-8749.1987.tb02482.x. PMID 3596065
- [Background] Eliasson AC, Krumlinde-Sundholm L, Rosblad B, Beckung E, Arner M, Ohrvall AM, Rosenbaum P. The Manual Ability Classification System (MACS) for children with cerebral palsy: scale development and evidence of validity and reliability. Dev Med Child Neurol. 2006 Jul;48(7):549-54. doi: 10.1017/S0012162206001162. PMID 16780622
- [Result] El-Shamy SM. Efficacy of Armeo(R) Robotic Therapy Versus Conventional Therapy on Upper Limb Function in Children With Hemiplegic Cerebral Palsy. Am J Phys Med Rehabil. 2018 Mar;97(3):164-169. doi: 10.1097/PHM.0000000000000852. PMID 29059068
- [Result] Gilliaux M, Renders A, Dispa D, Holvoet D, Sapin J, Dehez B, Detrembleur C, Lejeune TM, Stoquart G. Upper limb robot-assisted therapy in cerebral palsy: a single-blind randomized controlled trial. Neurorehabil Neural Repair. 2015 Feb;29(2):183-92. doi: 10.1177/1545968314541172. Epub 2014 Jul 11. PMID 25015650